CLINICAL TRIAL: NCT03219645
Title: A Randomized, Active-Controlled，Blinded-Endpoint and Parallel Group Pilot Trial Comparing the Antiplatelet Effects of Ginkgo Diterpene Lactone Meglumine Injection Plus Aspirin Versus Aspirin Alone in Patients With Acute Ischemic Stroke
Brief Title: Ginkgo Diterpene Lactone Meglumine Injection on Platelet Reactivity in Acute Ischemic Stroke
Acronym: GDPRS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Jiangsu Kanion Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-194（3）
Record Dates: First submitted 2017-07-05; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-05

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginkgo and aspirin (Active Comparator): Ginkgo Diterpene Lactone Meglumine Injection 25mg/5ml,once/day from Day 1 to Day 14. The injection must be added slowly into 0.9% sodium chloride injection and diluted to 250 ml , intravenous drip for about 2 hours;combined with Acetylsalicylic acid (Aspirin) given in a total dose of 300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 14.
  Interventions: Drug: Ginkgo Diterpene Lactone Meglumine Injection; Drug: Acetylsalicylic acid
- aspirin (Placebo Comparator): Acetylsalicylic acid (Aspirin) given in a total dose of 300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 14.
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Ginkgo Diterpene Lactone Meglumine Injection — The injection must be added slowly into 0.9% sodium chloride injection and diluted to 250 ml , intravenous drip for about 2 hours.
  Other Names: YinxingErtieneizhiPu'an Zhusheye
  Arms: Ginkgo and aspirin
Drug: Acetylsalicylic acid — Acetylsalicylic acid (Aspirin) given in a total dose of 300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 14.
  Other Names: Aspirin

SUMMARY:
This study evaluates the addition of Ginkgo Diterpene Lactone Meglumine Injection to aspirin in the treatment of acute ischemic stroke.Half of patient will receive Ginkgo Diterpene Lactone Meglumine Injection(25mg once/day D1-D14) and aspirin(300mg loading dose,then 100mg once/day D2-D14) in combination, while the other half will receive aspirin(300mg loading dose,then 100mg once/day D2-D14).

DETAILED DESCRIPTION:
The GDPRS trial is a prospective, randomized, single-centre, open-label, active-controlled, blinded-endpoint trial (a PROBE design concerning clinical trial). A total of approximately 40 patients (18 years≤Age≤ 80 years) with acute ischemic stroke (NIHSS < 12), who can be treated within 72 hours of symptom onset will be enrolled. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive a Ginkgo Diterpene Lactone Meglumine Injection 25mg/5ml,once/day from Day 1 to Day 14（the injection must be added slowly into 0.9% sodium chloride injection diluted to 250 ml , intravenous drip for about 2 hours）, combined with Acetylsalicylic acid (Aspirin) given in a total dose of 300 mg on the first day, followed by 100 mg once/day from Day 2 to Day 14. 2) the other group will receive a 300 mg loading dose of Aspirin on the day of randomization, followed by Aspirin 100 mg once/day from Day 2 to Day 14. The primary objective is to assess the anti-platelet effects of Ginkgo Diterpene Lactone Meglumine Injection combined with Aspirin versus Aspirin alone in patients with acute ischemic stroke. The study consists of 4 visits including the day of randomization, 24 hours after the first anti-platelet agents,Day 14±2days and Day 90±7days. The antiplatelet effects will be analyzed in total subjects. The trial is anticipated to complete in 6 months from the first subject recruitment , with 40 subjects recruited. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study. The trial has been approved by IRB(Institutional Review Board) /EC(Ethics Committee) in Renji hospital，Shanghai Jiaotong University School of Medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent;
2. Female or male with 18 years ≤age ≤ 80 years;
3. Within 72 hours symptom onset of ischemic stroke (diagnosis standard by the Chinese medical association of the fourth national conference on cerebrovascular disease);
4. Modified Rankin Scale Score ≤2 at the time of randomization;
5. NIHSS <12 points at the time of randomization;
6. Diagnosis of collaterals abstraction by phlegm and blood stasis in Traditional Chinese Medicine.

Exclusion Criteria:

1. Diagnosis of infection, cancer, autoimmune diseases,severe renal or hepatic insufficiency or deep vein thrombosis,etc;
2. Current treatment (last dose given within 10 days before randomization) with anticoagulation therapy or anti-platelet therapy;
3. Presumed cardiac source of embolus, e.g., atrial fibrillation, known prosthetic cardiac valves, suspected endocarditis or other cardioembolic pathology for stroke;
4. Low or high platelet count (<100 x10^9/L or >300 x10^9/L);
5. Clear indication for anticoagulation or thrombolysis;
6. Head imaging studies have confirmed that, encephalitis, brain tumor, brain abscess and cause similar symptoms of disease, or confirm with hemorrhagic cerebral infarction, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc;
7. Blood pressure elevated(systolic > 220mmHg or diastolic >120mmHg);
8. Pregnancy or lactation, and women of childbearing age not practicing reliable contraception who do not have a documented negative pregnancy test;
9. Known allergic to acetylsalicylic acid or Ginkgo Diterpene Lactone Meglumine;
10. With hemorrhagic disease or have a bleeding tendency;
11. Clear indication for Dual Antiplatelet Therapy with acetylsalicylic acid and clopidogrel;
12. Have to be fed through a nasal feeding tube;
13. Contraindication to acetylsalicylic acid;
14. Presumed probably poor adherence, or any other inappropriate conditions for patients to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
ARU on day 14 | 14 days
  Residual Platelet Reactivity defined as the value of Aspirin Reaction Unit (ARU) measured by VerifyNow® assay on day 14.

SECONDARY OUTCOMES:
PL-12 AA at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of acetylsalicylic acid.
PL-12 ADP at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of adenosine diphosphate.
PL-12 PAF at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®)using the inducer of PAF(Platelet activating factor).
PL-12 Coll at 24 hours and day 14 | 24hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®) using the inducer of collegen.
PL-12 Adr at 24 hours and day 14 | 24 hours,14 days
  Residual platelet reactivity detected by PL Platelet Analyser (SINNOWA®) using the inducer of adrenaline.
TEG-AA on day 14 | 14 days
  Residual platelet reactivity defined as the value of Maximum Amplitude- acetylsalicylic acid (MA-AA) measured by Thrombelastography Platelet Mapping Assay (TEG) using the inducer of acetylsalicylic acid.
TEG-ADP on day 14 | 14 days
  Residual platelet reactivity defined as the value of Maximum Amplitude- adenosine diphosphate (MA-AA) measured by Thrombelastography Platelet Mapping Assay (TEG) using the inducer of adenosine diphosphate
ARU at 24 hours | 24 hours
  Residual platelet reactivity defined as the value of Aspirin reaction unit (ARU) measured by VerifyNow® assay at 24 hours.
AA HOPR VerifyNow® | 24 hours，14 days
  High on-treatment platelet reactivity defined as Aspirin reactivity unit (ARU)> 555 measured by VerifyNow® assay.
Aspirinworks | 24 hours，14days
  Residual platelet reactivity detected by AspirinWorks.
Impairment | 14 days，90days
  Changes in NIHSS and mRS at 14 days and 90 days.
Modified Rankin Scale score changes | 14 days，90 days
  Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6
New vascular events defined as any event of the following: Any stroke (ischemic or hemorrhage). | 14 days
  All the new vascular events will be assessed by at least two neurologists based on neuroimaging and clinical feature. When there was disagreement, a third senior neurologist was consulted to reach a consensus decision.
New composite clinical vascular events (ischemic stroke/ hemorrhagic stroke/TIA/ myocardial infarction/ vascular death) as a cluster. | 14days，90 days
  The PLATO(Platelet Inhibition and Patient Outcomes) definition of fatal/life-threatening of major bleed is any one of the following: Fatal, Intracranial, Intrapericardial bleed with cardiac tamponade, Hypovolaemic shock or severe hypotension due to bleeding and requiring pressors or surgery, Clinically overt or apparent bleeding associated with a decrease in hemoglobin(Hb) of more than50 g/L, Transfusion of 4 or more units (whole blood or packed red blood cells [PRBCs]) for bleeding. The PLATO definition of other of major bleed is any one of the following:Significantly disabling (eg. intraocular with permanent vision loss), Clinically overt or apparent bleeding associated with a decrease in Hb of 30 g/L to 50 g/L, Transfusion of 2-3 units (whole blood or PRBCs) for bleeding.
Major bleed (PLATO definition), including fatal/life-threatening and other. | 14days，90 days
  The PLATO(Platelet Inhibition and Patient Outcomes) definition of fatal/life-threatening of major bleed is any one of the following: Fatal, Intracranial, Intrapericardial bleed with cardiac tamponade, Hypovolaemic shock or severe hypotension due to bleeding and requiring pressors or surgery, Clinically overt or apparent bleeding associated with a decrease in hemoglobin(Hb) of more than50 g/L, Transfusion of 4 or more units (whole blood or packed red blood cells [PRBCs]) for bleeding. The PLATO definition of other of major bleed is any one of the following:Significantly disabling (eg. intraocular with permanent vision loss), Clinically overt or apparent bleeding associated with a decrease in Hb of 30 g/L to 50 g/L, Transfusion of 2-3 units (whole blood or PRBCs) for bleeding.
Intracranial hemorrhagic events. | 14days，90 days
  Intracranial hemorrhagic events is assessed by brain computed tomography (CT) or gradient recalled echo (GRE) T2 star weighted MRI.
Total mortality. | 14days，90 days
  All deaths reported post-randomization will be recorded and adjudicated. Deaths will be subclassified by the adjudication committee as cardiovascular or non-cardiovascular.